CLINICAL TRIAL: NCT04075968
Title: The Effect of Cognitive Group Exercise Combined With Physical Exercise in Multiple Sclerosis Patients
Brief Title: The Effect of Cognitive Group Exercise Combined With Physical Exercise in MS
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstanbulPMRTRH
Record Dates: First submitted 2019-08-11; First posted 2019-09-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: exercise group; 6 weeks, twice a week, 30 minutes physical group exercises and 30 minutes general cognitive function exercises will be applied as groups.
  Interventions: Other: Cognitive exercise
- group 2: control group; patients will be given physical and cognitive home exercise program individually.
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Cognitive exercise — Cognitive exercise will be applied
  Groups: group 1
Other: Home exercise — Home exercise will be applied
  Groups: group 2

SUMMARY:
The aim of this study is to investigate the effect of cognitive rehabilitation in group with physical exercise in patients with Multiple Sclerosis. We assume that cognitive therapy is an effective treatment for multiple sclerosis.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of cognitive rehabilitation in group with physical exercise in patients with Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an Mini Mental State Test score less than 24
* Patients with an Extended Disability Status Scale score less than 4
* Patients trained for at least 5 years
* Patients who have not received steroid therapy in the last 1 month

Exclusion Criteria:

* Patients who have not passed at least 3 months from the last Multiple Sclerosis attack
* Patients with hearing and vision problems that may interfere with communication
* The patients who Have other neurological and psychiatric disorder that will cause cognitive impairment
* Patients receiving medical treatment for spasticity, tremor, bladder disorder and fatigue

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with definitive Multiple Sclerosis between 20-65 years, with an Mini Mental State Test score less than 24, with an Extended Disability Status Scale score less than 4, trained for at least 5 years, have not received steroid therapy in the last 1 month
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Neuro-psychometric Test (NPT) | 1 hour
  It is a test that evaluates memory, working memory, planning, organization, attendance span.Evaluation is made according to the number of items filled. The higher number items filled indicates the better status
Berg Balance Scale | 15 minutes
  It is a scale which consists of 14 items. Each item is scored on a five-point scale (0-4).The maximum score for this assessment is 56 and the minimum score for this assessment is 0. Scores below 45 indicate balance impairment. The higher point indicates the better status
Mini Mental State Test (MMST) | 10-15 minutes
  It is a test that evaluates different subset of cognitive status including attention, memory, language, orientation, visuospatial proficiency. It is scored on a scale of 0-30 with scores. Scores above 25 are interpreted as normal cognitive status.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | 3 minutes
  The MAS is a 6-point rating scale which assesses muscle tone by manually manipulating the joint through its available range of motion and clinically recording the resistance to passive movements. The lower point indicates the better status

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Esmeray, Study Chair — IstanbulPMHTRH
Locations (1):
- Health Sciences University Istanbul Physical Therapy and Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)